CLINICAL TRIAL: NCT00850759
Title: Using Virtual Reality to Train Children in Pedestrian Safety
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, David Schwebel, Professor of Psychology and Associate Dean for Research in the Sciences, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: F080715010; R01HD058573-01A1 (NIH)
Record Dates: First submitted 2009-02-24; First posted 2009-02-25 (Estimated); Results first posted 2013-11-20 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Street-crossing Ability; Pedestrian Safety
Keywords: pedestrian safety; street-crossing ability; road-crossing; children; injury prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- virtual reality (Experimental): street-crossing training in a virtual pedestrian environment
  Interventions: Device: virtual pedestrian environment
- computer and video (Active Comparator): exposure to training in pedestrian safety via computer software, internet games, and television videos
  Interventions: Device: computer and video
- streetside training (Active Comparator): one-on-one training in street-crossing skills by an adult, at a streetside location
  Interventions: Behavioral: streetside training
- no-contact control (No Intervention): no-contact control group.

INTERVENTIONS:
Device: virtual pedestrian environment — a computer-driven virtual pedestrian environment
  Arms: virtual reality
Device: computer and video — various computer-based and video-based programs such as Otto the Auto and WalkSafe
  Arms: computer and video
Behavioral: streetside training — one-on-one training by an adult with the child at streetside locations, to teach children street-crossing skills
  Arms: streetside training

SUMMARY:
Pedestrian injuries are among the leading causes of morbidity and mortality in American children ages 7-8, but existing behavior-oriented interventions achieve only modest success. One limitation to existing interventions is that they fail to provide children with the repeated practice needed to develop the complex perceptual and cognitive skills required for safe pedestrian activity.

Virtual reality (VR) offers a highly promising technique to train children in pedestrian safety skills. VR permits repeated unsupervised practice without risk of injury; automated feedback to children on success or failure in crossings; adjustment of traffic density and speed to match children's skill level; and an appealing and fun environment for training. The proposed research is designed to test the efficacy of virtual reality as a tool to train child pedestrians in safe street-crossing behavior.

A randomized controlled trial will be conducted with four equal-sized groups of children ages 7-8 (total N = 240). One group will receive training in an interactive and immersive virtual pedestrian environment. The virtual environment, already developed, has been demonstrated to have face, construct, and convergent validity. The second group will receive pedestrian safety training via video and computer strategies that are most widely used in American schools today. The third group will receive what is judged to be the most efficacious treatment currently available, individualized behavioral training at streetside locations. The fourth and final group will serve as a no-contact control group. All participants in all groups will be exposed to a range of field- and laboratory-based measures of pedestrian skill during baseline and post-intervention visits, as well as during a six-month follow-up assessment. Primary analyses will be conducted through linear mixed models designed to test change over time in the four intervention groups. We hypothesize all children in active learning groups will increase pedestrian safety skills, but the largest increase will be among children in the virtual reality group.

ELIGIBILITY:
Inclusion Criteria:

* 7 and 8 year old children living in Birmingham, Alabama, area

Exclusion Criteria:

* family plans to move within 6 months of recruitment
* visual or perceptual impairment (e.g., blindness) that are uncorrected and would prevent valid participation in protocol
* physical impairment (e.g., use of wheelchair) that would prevent valid participation in protocol
* cognitive impairment (e.g., moderate mental retardation) that would prevent valid participation in protocol

Ages: 7 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2009-10; Primary Completion 2012-05 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C Schwebel, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Youth Safety Lab, University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Background] Schwebel DC, McClure LA. Using virtual reality to train children in safe street-crossing skills. Inj Prev. 2010 Feb;16(1):e1-5. doi: 10.1136/ip.2009.025288. PMID 20179024
- [Background] Schwebel DC, Davis AL, O'Neal EE. Child Pedestrian Injury: A Review of Behavioral Risks and Preventive Strategies. Am J Lifestyle Med. 2012 Jul;6(4):292-302. doi: 10.1177/0885066611404876. Epub 2011 Jun 17. PMID 23066380

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment from a variety of community sources between October 2009 and September 2011
Pre-assignment Details: 9 excluded prior to group assignment, for these reasons: Not meeting inclusion criteria; child of incorrect age (n = 3) Not meeting inclusion criteria; child unable to understand protocol (n = 3) Did not complete baseline assessment (n = 3)
Period: Overall Study
Arm/Group | Virtual Reality | Computer and Video | Streetside Training | No-contact Control
Started | 59 | 57 | 57 | 58
Completed | 52 | 52 | 52 | 55
Not Completed | 7 | 5 | 5 | 3
Not completed — Lost to Follow-up | 7 | 5 | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Virtual Reality | Computer and Video | Streetside Training | No-contact Control | Total
Number analyzed (Participants) | 59 | 57 | 57 | 58 | 231
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 59 | 57 | 57 | 58 | 231
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.9 (0.67) | 8.1 (0.63) | 7.9 (0.68) | 8.1 (0.63) | 8.0 (0.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 35 | 35 | 30 | 132
  Male | 27 | 22 | 22 | 28 | 99
Region of Enrollment [Number; unit: participants]
  United States | 59 | 57 | 57 | 58 | 231

OUTCOME MEASURES:

1. Primary Outcome: Street-crossing Ability
Description: average count of hits/close calls per participant in virtual environment, out of 30 crossings
Time Frame: post-training and again 6 months later
Measure: Mean (Standard Deviation); unit: number of hits/close calls
Arm/Group | Virtual Reality | Streetside Training | Computer and Video | No-contact Control
Number analyzed (Participants) | 52 | 52 | 52 | 55
number of hits/close calls
  post-intervention hits/close calls in VR | 2.7 (1.6) | 2.3 (1.2) | 2.6 (1.6) | 3.0 (1.6)
  6 month follow-up hits/close calls in VR | 2.1 (1.4) | 1.7 (1.1) | 2.3 (1.5) | 2.6 (1.6)
Statistical Analysis 1: Comparison: Virtual Reality vs Streetside Training vs Computer and Video vs No-contact Control; Test type: Superiority or Other; p < 0.05, ANOVA; Slope = 0.04

ADVERSE EVENTS:
Description: Both serious and other (non-serious) adverse events were collected and assessed, but non were observed.
Arm/Group | Virtual Reality | Computer and Video | Streetside Training | No-contact Control
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/57 | 0/57 | 0/58
Other Adverse Events (participants affected / at risk) | 0/59 | 0/57 | 0/57 | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No